CLINICAL TRIAL: NCT01100333
Title: Observational Study GONAL-f® Consort
Brief Title: GONAL-f CONSORT (Consistency in r-hFSH Starting Doses for Individualised Treatment)
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: 700623-500
Record Dates: First submitted 2010-02-24; First posted 2010-04-08 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2013-01

CONDITIONS: Infertility
Keywords: Infertility; Reproductive technologies, Assisted; r-hFSH; Gonal-f
MeSH Terms: conditions — Infertility; Helping Behavior | interventions — Glycoprotein Hormones, alpha Subunit; follitropin alfa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole Blood

INTERVENTIONS:
Drug: Recombinant human follicle stimulating hormone (r-hFSH) — Recombinant hFSH prescribed according to prescriber's judgement
  Other Names: Gonal-f

SUMMARY:
This non-interventional study (NIS) is planned to examine the consistency of the dose recommended by the doctor for the first stimulation day with the dose recommended by the CONSORT calculator.

DETAILED DESCRIPTION:
Since the introduction of the first recombinant human follicle stimulating hormone (FSH) preparation Gonal-f in the year 1996, a pure drug is available as raw material, which is independent of human urine due to biotechnological methods and consequently can be produced free of contaminating proteins. In accordance with the recommendations of European Medicines Agency (EMEA) in February 1999, on the basis of data from clinical studies, Gonal-f should be regarded as the more effective preparation in comparison to urinary FSH. Serono has developed a dose calculator, the CONSORT calculator, after analyzing the data from clinical studies for Gonal-f. This non-interventional study is planned to examine the consistency of the dose recommended by the doctor for the first stimulation day with the dose recommended by the CONSORT calculator. All subjects, who undergo stimulation with Gonal-f in preparation for a technology of the assisted conception in accordance with the permitted indication, will be included in this non-interventional study.

OBJECTIVES

Primary Objective:

* To examine, how far the dose recommended by the doctor for the first stimulation day varies from the dose recommended by the CONSORT calculator

ELIGIBILITY:
Inclusion Criteria:

* Female subjects undergoing stimulation with Gonal-f in ART in accordance with the permitted indication
* Subjects below 35 years of age
* Subjects who have a Body mass index below 30
* Subjects with a basal FSH below 12 I.E./l and is downregulated in the long gonadotropin hormone releasing hormone agonist (GnRHa) Protocol

Max Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects undergoing Assisted Reproductive Technologies (ART) receiving Gonal-f in Germany
Sampling Method: Probability Sample
Enrollment: 2552 (Actual)
Dates: Start 2008-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Consistency of dose of Gonal-f recommended by the doctor for the first stimulation day with the dose recommended by the CONSORT calculator | 6 month

SECONDARY OUTCOMES:
Efficacy parameters | 6 month
  Total dose and the necessity of a dose adjustment during stimulation period, number of the obtained ova after hCG administration, the duration of the stimulation,stimulation dose on the last stimulation day

CONTACTS AND LOCATIONS:
Overall Officials: W. Bilger, Study Chair — Merck Serono GmbH, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Universitätsmedizin Charitè Berlin, Schumann Straße 20/21, Berlin, State of Berlin, Germany